CLINICAL TRIAL: NCT05895903
Title: Evaluation of Dental Implant Stability in Narrow Alveolar Ridges Utilizing Osseodensification Technique Versus Screw Expansion: A Comparative Clinical Study
Brief Title: Alveolar Ridges Expansion Using Osseodensification Versus Screw Expansion Technique
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Baghdad (Other)
Responsible Party: Principal Investigator, Nawfal Hasan Abbas Tofan, principal investigator, University of Baghdad
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: 07718814
Record Dates: First submitted 2023-05-15; First posted 2023-06-09 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-05

CONDITIONS: Dental Implant Failed; Bone Fracture; Bone Infection
Keywords: Dental implant stability; narrow alveolar ridges; alveolar ridge expansion
MeSH Terms: conditions — Fractures, Bone

STUDY DESIGN:
Intervention Model Description: Nineteen patients (12 females and 7 males) with narrow alveolar ridges participated in this research. Forty-six osteotomy sites were prepared, and 41 DIs were installed. A randomized allocation sequence created using GraphPad Prism 9 software divided the patients in two groups. The SE technique group consisted of 21 DIs after alveolar bone expansion with threaded screw expander drills, and the OD group consisted of 20 DIs after alveolar ridge expansion with Densah® burs.
Who Masked: Participant, Care Provider, Investigator
Masking Description: A randomized allocation sequence created using GraphPad Prism 9 software divided the patients in two groups.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Screw expansion group (Active Comparator): threadform screw expanders with special condensing burs for lateralization and compaction of bone while simultaneously placing dental implants
  Interventions: Device: Screw expander
- Osseodensification group (Active Comparator): special drills to expand narrow alveolar ridges.These drills share similar advantages with osteotomes in terms of greater tactile sensitivity, faster speed, and low heat generation, all of which help to maintain healthy bone and enhance implant osseointegration.
  Interventions: Device: Osseodensification drills

INTERVENTIONS:
Device: Screw expander — threadform screw expanders with special condensing burs for lateralization and compaction of bone
  Other Names: Threads expander
  Arms: Screw expansion group
Device: Osseodensification drills — special drills to expand narrow alveolar ridges.
  Other Names: Densah burs
  Arms: Osseodensification group

SUMMARY:
Alveolar ridge expansion is suggested for alveolar crest thicknesses of 3-5 mm. Osseodensification (OD) and screw expansion (SE) techniques have been utilized to expand narrow alveolar ridges (NAR). This study aims to compare the implant stability quotient (ISQ) values of endosteal dental implants (DIs) inserted into NAR via osseodensification versus manual screw expansion.

DETAILED DESCRIPTION:
This study aimed to evaluate implant primary stability using Densah bur in comparison with screw expander in narrow alveolar ridge.

The patient is instructed to gargle with 0.2% chlorhexidine mouthwash, scrubbing the perioral area with 10% povidone iodine and draping the patient head with disposable drapes.

The surgery will be performed under local anesthesia using lidocaine hydrochloride 2% with adrenaline 1:8000, the surgical procedure started with flap reflection. A mucoperiosteal elevator was used to reflect the buccal and palatal flaps that were enough to expose the crestal part of alveolar ridge with clear visibility and accessibility.

For Expander group:

The screw expanders will be use to expand the osteotomy site. The diameters will be use 2.3mm ,2.6 mm, 3 mm, 3.4 mm, 3.8 mm in a successive manner. Each expander will be screw until 10 mm of depth is reached as mark on the expander. Each expanders is gently screwed half turn at a time; to allow slow and gradual expansion of the bone . When necessary, the kit ratchet is used to reach the full depth required. After the use of the final expander, an implant of appropriate size will place.

FOR DENSAH BUR GROUP :

The Implant motor is set in an anti-clockwise direction and drilling speed is set at 1000 rpm. Densah Burs will use in increasing diameters of 2mm,2.3mm,2.5 mm, 3.0 mm,3.3mm, and 3.5 mm in asuccessive manner and under copious irrigation with sterile saline.

When the haptic feedback of the bur is encountered, pressure is modulated by a pumping motion in and out of the osteotomy until 10mm of depth is reached as mark on the bur . After the use of the final expander, an implant of appropriate size will place.

For both groups After implant placement, the integrity of the buccal bone will examine for any cracks. The Smart peg* corresponding with the implant system is placed on the implant and Osstell device is use to measure ISQ from buccal, lingual, mesial, and distal directions. For each side, three reading were taken and an average was calculated. A healing collar will place on the implant, then the flap will approximate and suture around healing collar.

Patients is instruct to take an antibiotic after surgery every 24 hours for a week and to start non-steriodal anti-inflammatory drug every 8 hours for 2-3 days; to control the possible post operative pain and edema. Antiseptic mouthwash is also continue 3 times daily for 14 days. The patients will informe with the next appointment date so that the sutures are to be removed after 1 week.

ELIGIBILITY:
1. Patient's age ≥18 years.
2. Absence of any medical disease that compromise wound healing.
3. patient with good oral hygiene.
4. Narrow alveolar ridge (2,5-5 mm) and the period after tooth extraction is at least 6 months.

Exclusion Criteria:

* 1. Uncontrolled medically compromised patients. 2. Heavy smokers (> 20 cigarettes per day) 3. Patient with parafunctional habits. 4. Local infection at implant site.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2021-12-15 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2023-01-02 (Actual)

PRIMARY OUTCOMES:
Primary stability | At the time of surgery
  After implant insertion, the multipeg was screwed into the implant fixture, and stability measurement was conducted with the Osstell® ISQ device in two directions (buccolingual and mesiodistal). The mean of these two measurements was recorded as an ISQ value.
Alveolar ridge thickness | At the time of surgery
  Alveolar bone thickness was measured after osteotomy site preparation.

SECONDARY OUTCOMES:
secondary stability | 6 months
  After implant insertion, the multipeg was screwed into the implant fixture, and stability measurement was conducted with the Osstell® ISQ device in two directions (buccolingual and mesiodistal). The mean of these two measurements was recorded as an ISQ value.

CONTACTS AND LOCATIONS:
Overall Officials: NAWFAL HASAN ABBAS, B.D.S, Principal Investigator — Baghdad university/College of Dentistry
Locations (1):
- college of dentistry/University of Baghdad, Baghdad, Iraq